CLINICAL TRIAL: NCT04967521
Title: SARC041: Phase 3 Randomized Double-Blind Study of Abemaciclib Versus Placebo in Patients with Advanced Dedifferentiated Liposarcoma
Brief Title: SARC041: Study of Abemaciclib Versus Placebo in Patients with Advanced Dedifferentiated Liposarcoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SARC041
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Advanced Dedifferentiated Liposarcoma
MeSH Terms: interventions — abemaciclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abemaciclib (Experimental): Abemaciclib will be administered 200mg orally twice a day. Each cycle is 28 days.
  Interventions: Drug: Abemaciclib
- Placebo Arm (Placebo Comparator): Patients will be randomized 1:1 and will receive placebo if they are randomized to the placebo arm of the study. Each cycle is 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib will be administered 200mg orally twice a day. Each cycle is 28 days.
  Other Names: LY2835219
  Arms: Abemaciclib
Drug: Placebo — Placebo will be administered orally twice a day. Each cycle is 28 days.
  Arms: Placebo Arm

SUMMARY:
This is a Phase 3 randomized double-blind study of abemaciclib versus placebo. Patients with progression of disease will cross over to open label abemaciclib.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled study of patients with advanced, recurrent and/or metastatic DDLS.

Patients will be randomized 1:1 between abemaciclib and placebo and followed for disease progression. For those patients with progression of disease (by RECIST) on placebo, crossover to active drug will be offered to patients if they remain eligible for the clinical trial in all other respects. Unblinding and crossover is only allowed for radiographic progression (not clinical progression). Real-time radiology review by the treating physician will allow for rapid crossover for patients with progression on placebo. If patients are deemed to have disease that is too rapidly progressive to be considered for a randomized, double-blind, placebo-controlled clinical trial, they should be excluded from consideration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of dedifferentiated liposarcoma which is locally recurrent and/or metastatic. This study will accept the diagnosis made at the investigator's center.
* ECOG Performance Status of 0 or 1.
* At least one site of measurable disease on CT/MRI scan as defined by RECIST 1.1 criteria. Baseline imaging must be performed within 28 days of Day 1 of study.
* Adequate organ function
* The patient can swallow oral medications.
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the patient did not receive radiotherapy).
* Written, voluntary informed consent
* Fertile men and women of childbearing potential must agree to use a highly effective method of birth control during the treatment period and for 3 weeks after last study drug administration in both sexes. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ seven days of the first dose of abemaciclib.
* Highly effective methods of birth control include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.
* Measurable disease and evidence of progression of disease as defined by RECIST 1.1 (including newly diagnosed disease, new disease sites in a patient who was previously NED, or a 20% growth of existing lesions within 6 months of registration).
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery within 3 months from completion of therapy to sites of CNS metastatic disease and are without evidence of clinical progression.

Exclusion Criteria:

* Patients with documentation of well-differentiated liposarcoma only are specifically excluded, owing to its characteristically slow growth. If high grade areas are suspected (dedifferentiation), but not proved by pathology analysis (e.g. after primary resection of a well-differentiated liposarcoma), a biopsy must be performed to demonstrate the high-grade dedifferentiated disease. If there is a question regarding the diagnosis, the PI should be consulted.
* Patients with bulky disease who urgently need cytotoxic chemotherapy (likely with doxorubicin + ifosfamide) will be excluded from this study. This is determined by the treating physician. If there is a question regarding the appropriateness of the patient for enrollment, the PI should be consulted.
* Prior systemic therapy with abemaciclib or any other selective CDK4 inhibitor (such as palbociclib)
* Concurrent, clinically significant, active malignancies within 12 months of study enrollment
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery within 3 weeks prior to Day 1 of study or who have not recovered adequately from prior surgery
* Patients with resectable for curative intent disease
* Patients that have GI absorption disorders that would impact the administration of oral abemaciclib.
* Women who are pregnant or nursing/breastfeeding.
* Known hypersensitivity to abemaciclib.
* Patients with untreated central nervous system disease.
* Inability to comply with protocol required procedures
* Patients currently taking the following drugs may interact with abemaciclib. Please refer to Section 5.2 of protocol.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the progression-free survival of patients treated with abemaciclib versus placebo | 5 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
To determine the objective response rate by RECIST 1.1 | 5 years
  A patient will be deemed to have an objective response if they have a confirmed complete response or partial response as determined by RECIST v1.1
To determine PFS after crossover for patients initially randomized to placebo | 5 years
  PFS after crossover will only be determined for patients who were randomized to placebo. It will be measured from the start of abemaciclib treatment until the occurrence of disease progression or death due to any cause prior to documented disease progression.
To determine overall survival | 5 years
  The length of time from the start of treatment that patients diagnosed with sarcoma are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dickson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Colorado Cancer Center, Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No